CLINICAL TRIAL: NCT04048980
Title: Care of Older People With Cognitive Impairment or Dementia Hospitalized in Traumatology Units
Acronym: CARExDEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Puerta de Hierro University Hospital (Other); Hospital Universitario Marqués de Valdecilla (Other); Complejo Hospitalario de Navarra (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Adelaida Zabalegui Yarnoz, Subdirector Reasearch and Education in Nursing, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2017/0499
Record Dates: First submitted 2019-07-26; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Dementia; Femur Fracture; Continuity of Patient Care
Keywords: intervention; elderly; nursing care
MeSH Terms: conditions — Dementia; Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients with dementia or cognitive impairment and femur fracture receiving the traditional care in traumatology units.
- Experimental Group (Experimental): Patients with dementia or cognitive impairment and femur fracture receiving an intervention in traumatology units.
  Interventions: Behavioral: CARExDEM

INTERVENTIONS:
Behavioral: CARExDEM — CARExDEM is an educational program addressed to nurses working in traumatology units and looking after patients with dementia. This intervention pretends to provide strategies to nurses for cognitive impairment management in acute hospital settings, to raise awareness about personalized care in dementia and to improve continuity of care in acute situations in PwD. Training sessions will be held to inform and train nurses about care of PwD and their caregivers by the research team in each hospital.
  Arms: Experimental Group

SUMMARY:
This is a quasi-experimental design with repeated observations, taken at baseline, post-intervention, and at one and three months post-intervention. Participants will be patients hospitalized with cognitive disorders o dementia and a femur fracture. The study will be developed in four general hospitals in Spain and will include 430 patients with dementia (PwD) and their informal caregivers (IC). The study sample will be assigned to the control group (n=215) from each hospital involved and will receive the standard treatment. After completing the recruitment for the control group, the investigators will start to recruit patients until experimental patient group is complete (n=215) from each hospital to whom the CARExDEM intervention will be implemented.

DETAILED DESCRIPTION:
The high vulnerability of PwD hospitalized generates the need to confront this challenge from a global and continuous perspective along with the clear lack of intervention studies with PwD hospitalized at a national and international level.

The aim of this study is to design, implement and evaluate the effectiveness of an intervention program for nurses looking after hospitalized patients with proximal femur fracture and dementia or cognitive impairment, in acute hospitals and its impact in quality of care, morbidity reduction, improvement of continuity of care and reduction in costs.

The study will be conducted in four traumatology units of high technology public hospitals across Spain: the autonomous communities included are Catalonia (Hospital Clinic Barcelona), Madrid (Hospital Puerta de Hierro Madrid), Cantabria (Hospital Marqués de Valdecilla) and Navarra (Complejo hospitalario de Navarra). The study will be held in a 3 year frame time.

Participants will be patients with dementia and their caregiver elected consecutively (n=432), and healthcare professionals working in the traumatology unit. All questionnaires selected are valid and reliable and widely used among studies with PwD. All questionnaires were translated already to Spanish and we have permission of the authors for using them. They are structured in Likert scaling. The whole questionnaire can be completed in 45 minutes (for patient questions) and 15 minutes (for informal caregivers).

Data will be collected by trained interviewers at hospital admission (within 24 hours), discharge, 1 moth follow up at the outpatient traumatology visit and 3 months follow up (phone call). Questionnaires have been customized in one document according to the collection phase. Questions will be responded according to patient and caregiver data.

Procedure

The study will be conducted in 3 phases:

1. Pre-intervention stage: Program design Design of the intervention CARExDEM: It will be developed from the results obtained from the European study RightTimePlaceCare. They evaluated care of PwD and their caregivers in Europe using the Balance of Care methodology. This method implies expert healthcare professionals (nurses, physicians, physiotherapists, social workers and care assistants) in care of patients with dementia or cognitive impairment and traumatology. The experts will reach a consensus about the best care needed under these circumstances, constituting the educational intervention CARExDEM.

   CARExDEM is an educational program aimed for nurses and other health professionals looking after PwD and a femur fracture. Information and dynamic educational sessions will be adapted from clinical guidelines and best practices. This intervention pretends to provide nurses with strategies in the management of PwD in acute care and to raise awareness about the importance on individualized care in these patients to improve continuity of care in exacerbated situations on PwD.

   Educational training will be held, approved by unit managers and the research team, and all hospitals will follow the same protocol. The investigators will train nurses about the care guide including aspects such as use of physical restraints, psychotropic medication, falls, functional capacity and pain.
2. Implementation of the intervention CARExDEM A pilot test will be monitored prior to implementation in each hospital. The investigators will consider opinions of experts and informal caregivers related to its applicability, follow up, population participation and time cost/savings. Once the intervention is implemented, the investigators will follow closely in case of doubts or barriers. Weekly meetings will be held to review the nurses training.
3. Follow up and evaluation of the CARExDEM implementation related to costs Data will be introduced in a database and results will be evaluated by an expert statistician. The research team will discuss the results and outcomes will be presented in Congresses and articles.

Intervention The intervention will be designed following the Balance of Care (BoC) methodology. This methodology implies multidisciplinary experts (nurses, physicians, physiotherapists, social workers and care assistants) evaluating resources and activities needed for an optimum care of PwD admitted to traumatology units.

CARExDEM is an educational program addressed to nurses working in traumatology units and looking after patients with dementia. The intervention will be complemented with a checklist guide that will enhance implication and raise awareness when implementing it. Information and dynamics of training sessions will be adapted according to clinical guidelines and best practice.

Statistical Analysis Descriptive analysis will be used for baseline data. Categorical variables will be represented with absolute frequencies and percentages. For continuous variables, mean values, standard deviation or medians will be calculated. To study the effect of the intervention, analysis of co-variance will be approached (ANCOVA), also Student's t-test in continuous variables and McNemar test in categorical variables. Sensibility will be analyzed to compare basal data of participants finishing the study and those who will not finish it. Outcomes measured will evaluate longitudinal changes from all the collection phases; baseline (admission), discharge, 1 month and 3 months follow up. Data from the four hospitals participating in the study also will be compared according to own resources. Confidence intervals of 95% will be calculated. Values of p< 0,05 will be considered significant. Confidence interval of 95% will be calculated. Statistical analysis will be done with R program, 3.2.3. Version for Windows. The research team will reflect about the analyzed data and will issue a final report including the CARExDEM program with the required modifications identified following the implementation evaluation. This will ease the implementation of the program in other hospitals subsequently.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 65

   * Hospitalized for surgery
   * Informal caregiver able to understand the recommendations of health professionals
   * Score of 5 or less in the Short Portable Mental Status Questionnaire (SPMSQ) test
   * Signed informed consent form.
2. Informal caregivers:

   * Living with the PwD or visiting at least three times per week at home or nursing home
   * Signed informed consent form.

Exclusion Criteria:

* Patients younger than 65
* Psychiatric symptoms or Korsakov syndrome
* No signed consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of Restraints | 3 months
  Adapted questionnaire from Hammers et al. 8 items (Never - more tan once a day).7 items where each ítem is a type of restraint: Belt, chair or wheelchair with blockages (tables), handrails, adjusts sheets, infrared, sensors,door blockage in room.There is no total scoring, as items will be assessed individually to identify the type of restraint used.
Psychotropic medication | 3 months
  Records on chart about use of psychotropic medication. Name of medication administered during hospitalization or at home.
Pain assessment in dementia: MPAINAD scale | 3 months
  PAINAD scale (Pain assessment in dementia). 5 items evaluating breathing, negative vocalization, facial expression, body language and consolability. The total score ranges from 0-10 points. A possible interpretation of score is: 1-3=mild pain, 4-6=moderate pain, 7-10=severe pain
Falls (number) | 3 months
  Record from proxy if any falls (witnessed/unwitnessed) It is considered a fall when a patient reached the floor from another level. Number of falls recorded
Functional capacity | 3 months
  Barthel Index: 10 items evaluating physical impairment; where each item scores 0-15 depending on item (0=dependent, 15 independent). Several authors have proposed guidelines for interpreting Barthel scores. Shah et al. suggested that scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency. Total scoring Katz Index: 6 items. Evaluating activities by dependence or Independence. Scoring ranges from 0-6 where 0 is Low (patient very dependent and 6 High, patient very independent)
Knowledge of nurses | 3 months
  An "ad hoc" questionnaire was created to know the nurses knowledge of care of patients with dementia. Sociodemographic data as age, level of studies, experience in years at the hospital, and questions about self-assessment abilities,implication with patient care, patient empowerment, evaluation of self training. The questionnaire has 25 questions and applies from (all patients to no patients). It also has open questions about barriers and facilitators regarding patient education in the unit. There is no total scoring, as questions are qualitative mostly and it not considered a scale.
Informal Caregiver Costs | 3 months
  RUD (Resource Utilization in Dementia) questionnaire. Evaluates the caregiver's input on resource utilization. Frequency and duration of hospitalization, visits to health care professionals and type of care, medication use, use of social services, caregiver time spent with patient on basic activities and instrumental activities of daily living, caregiver work status and whether informal caregiver substitutes for paid work. Time (in hours) of dedication of informal caregiver for patient. Healthcare services used in the last month (primary care doctor or nurse, physiotherapists, social services...) There is no total scoring as it is not a scale. Costs will be estimated by multiplying the number of units for each relevant factor from the questionnaire with the corresponding unit price vector. Total costs will be measured as average monthly costs in euros.
Caregiver burden | 3 months
  CRA (Caregiver reaction assessment) a 24-item instrument designed to measure the reactions of family members to caring for elderly relatives with a variety of illnesses. Items are rated on a 5-point scale (from "strongly agree" to "strongly disagree"). Caregiver's esteem (7 items);Lack of family support (5 items);Impact on finances assesses the adequacy, difficulty, and strain of finances on the caregiver and family (3 items);Impact on schedule (5 items);Impact on health assesses the caregiver's capability to provide care and health in relation to caregiving (4 items).Burden related to disrupted time (range 5-25), financial problems (range 3-15), lack of family support (range 5-25), health problems (range 4-20), and self-esteem (range 7-35). Higher=worse (greater burden)
Cognitive status | 3 months
  NPI-Q (Neuro-psychiatric inventory). 12 items evaluating psychopathology in dementia.
  Severity
  1. = Mild (noticeable, but not a significant change)
  2. = Moderate (significant, but not a dramatic change)
  3. = Severe (very marked or prominent; a dramatic change). Scoring for distress: 0 = Not distressing at all Distress
  0 = Not distressing at all
  1. = Minimal (slightly distressing, not a problem to cope with)
  2. = Mild (not very distressing, generally easy to cope with)
  3. = Moderate (fairly distressing, not always easy to cope with)
  4. = Severe (very distressing, difficult to cope with)
  5. = Extreme or very severe (extremely distressing, unable to cope with). Total score: After all domains have been scored, adding up the total score out of a possible 144. (Less tan 20=mild problem, 20-50= moderate disturbance, 50+=severe disturbance
Comorbidity | 3 months
  Charlson comorbidity index (19 items) evaluating comorbidity. Comorbid diseases were coded as: 0=absent; 1=present. Severity was coded as: 1=not ill; 2=mildly ill; 3=moderately ill; 3=severely ill and 5=moribund. To create a scoring, the method Hutchinson and Thomas combining age and comorbidity.

SECONDARY OUTCOMES:
Psychotropic medication administration | 3 months
  Records on chart about use of psychotropic medication. Dose (mg) during hospitalization or at home.
Frequency on psychotropic medication | 3 months
  Records on chart about use of psychotropic medication. Frequency (calculated in 24h) during hospitalization or at home
Injuries related to falls | 3 months
  Record from proxy if any falls (witnessed/unwitnessed) It is considered a fall when a patient reached the floor from another level. Injuries like bruises, open wounds, luxation or fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Risco E, Zabalegui A, Miguel S, Farre M, Alvira C, Cabrera E. [Application of the Balance of Care model in decision-making regarding the best care for patients with dementia]. Gac Sanit. 2017 Nov-Dec;31(6):518-523. doi: 10.1016/j.gaceta.2016.07.006. Epub 2016 Oct 15. Spanish. PMID 27751643
- [Background] Mosk CA, Mus M, Vroemen JP, van der Ploeg T, Vos DI, Elmans LH, van der Laan L. Dementia and delirium, the outcomes in elderly hip fracture patients. Clin Interv Aging. 2017 Mar 10;12:421-430. doi: 10.2147/CIA.S115945. eCollection 2017. PMID 28331300
- [Background] Farre M, Haro JM, Kostov B, Alvira C, Risco E, Miguel S, Cabrera E, Zabalegui A. Direct and indirect costs and resource use in dementia care: A cross-sectional study in patients living at home. Int J Nurs Stud. 2016 Mar;55:39-49. doi: 10.1016/j.ijnurstu.2015.10.012. Epub 2015 Nov 19. PMID 26632506
- [Background] Briggs R, Dyer A, Nabeel S, Collins R, Doherty J, Coughlan T, O'Neill D, Kennelly SP. Dementia in the acute hospital: the prevalence and clinical outcomes of acutely unwell patients with dementia. QJM. 2017 Jan;110(1):33-37. doi: 10.1093/qjmed/hcw114. Epub 2016 Aug 2. PMID 27486262
- [Background] Foebel AD, Liperoti R, Onder G, Finne-Soveri H, Henrard JC, Lukas A, Denkinger MD, Gambassi G, Bernabei R; SHELTER Study Investigators. Use of antipsychotic drugs among residents with dementia in European long-term care facilities: results from the SHELTER study. J Am Med Dir Assoc. 2014 Dec;15(12):911-7. doi: 10.1016/j.jamda.2014.07.012. Epub 2014 Sep 24. PMID 25262195
- [Background] Verbeek H, Meyer G, Leino-Kilpi H, Zabalegui A, Hallberg IR, Saks K, Soto ME, Challis D, Sauerland D, Hamers JP; RightTimePlaceCare Consortium. A European study investigating patterns of transition from home care towards institutional dementia care: the protocol of a RightTimePlaceCare study. BMC Public Health. 2012 Jan 23;12:68. doi: 10.1186/1471-2458-12-68. PMID 22269343
- [Background] Johansson Stark A, Charalambous A, Istomina N, Salantera S, Sigurdardottir AK, Sourtzi P, Valkeapaa K, Zabalegui A, Bachrach-Lindstrom M. The quality of recovery on discharge from hospital, a comparison between patients undergoing hip and knee replacement - a European study. J Clin Nurs. 2016 Sep;25(17-18):2489-501. doi: 10.1111/jocn.13278. Epub 2016 Jun 6. PMID 27264877
- [Background] Librero J, Peiro S, Ordinana R. Chronic comorbidity and outcomes of hospital care: length of stay, mortality, and readmission at 30 and 365 days. J Clin Epidemiol. 1999 Mar;52(3):171-9. doi: 10.1016/s0895-4356(98)00160-7. PMID 10210233
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Warden V, Hurley AC, Volicer L. Development and psychometric evaluation of the Pain Assessment in Advanced Dementia (PAINAD) scale. J Am Med Dir Assoc. 2003 Jan-Feb;4(1):9-15. doi: 10.1097/01.JAM.0000043422.31640.F7. PMID 12807591
- [Background] Given CW, Given B, Stommel M, Collins C, King S, Franklin S. The caregiver reaction assessment (CRA) for caregivers to persons with chronic physical and mental impairments. Res Nurs Health. 1992 Aug;15(4):271-83. doi: 10.1002/nur.4770150406. PMID 1386680
- [Background] Mira JJ, Nuno-Solinis R, Guilabert-Mora M, Solas-Gaspar O, Fernandez-Cano P, Gonzalez-Mestre MA, Contel JC, Del Rio-Camara M. Development and Validation of an Instrument for Assessing Patient Experience of Chronic Illness Care. Int J Integr Care. 2016 Aug 31;16(3):13. doi: 10.5334/ijic.2443. PMID 28435422
- [Background] Wimo A, Wetterholm AL, Mastey V, Winblad B. Evaluation of the resource utilization and caregiver time in Anti-dementia drug trials - a quantitative battery. in: Wimo A, Karlsson G, Jönsson B, Winblad B (eds) . The Health Economics of Dementia, 1998. Wiley's, London, UK
- [Background] Abellán A, Pujol R. Un perfil de las personas mayores en España. Indicadores estadísticos básicos. 2016. Consejo Superior de Investigaciones Científicas (CSIC). Centro de Ciencias Humanas y Sociales (CCHS). Envejecimiento en red.
- [Derived] Casafont C, Risco E, Piazuelo M, Ancin-Pagoto M, Cobo-Sanchez JL, Solis-Munoz M, Zabalegui A. Care of older people with Cognitive Impairment or Dementia Hospitalized in Traumatology Units (CARExDEM): a quasi-experiment. BMC Geriatr. 2020 Jul 16;20(1):246. doi: 10.1186/s12877-020-01633-5. PMID 32677894